CLINICAL TRIAL: NCT04444726
Title: Phototherpy Versus Tap Water Iontophoresis for Management of Atopic Dermatitis in Children, Randomized Clinical Trial.
Brief Title: Phototherpy Versus Tapwater Iontophoresis for Management of Atopic Dermatitis in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Ibrahim Ali, Assistant Professor , department of physical therapy for basic science, Faculty of Physical Therapy , Cairo university., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2776
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, Phototherapy, iontophoresis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phototherapy "PUVA" +traditional medical treatmentn (Experimental): patient sock his hands in a bath containing water with the constitution of psoralen "meladinine " capsule for 20 minutes then irradiated at the UVA device for 3 sessions per week for 8 weeks Plus the traditional medical treatment. which is the betamethasone dipropionate 0.05% " diprolene for 2 times a day for 8 weeks.
  Interventions: Device: Ultra Violet A Device.+ Topical medical treatment; Drug: Topical medical treatment (Betamethasone dipropionate 0.05% " diprolene " )
- Tap Water Iontophoresis + Traditional medical treatment (Experimental): Tap-water iontophoresis was given 3 times weekly for 10 min The direct current level was slowly increased, guided by the occurrence of tingling sensations. The maximum level was 30mA. Plus the traditional medical treatment. which is the betamethasone dipropionate 0.05% " diprolene for 2 times a day for 8 weeks.
  Interventions: Device: Iontophoresis device + Topical medical treatment; Drug: Topical medical treatment (Betamethasone dipropionate 0.05% " diprolene " )
- traditional medical treatment (Active Comparator): Traditional medical treatment. which is the betamethasone dipropionate 0.05% " diprolene for 2 times a day for 8 weeks.
  Interventions: Drug: Topical medical treatment (Betamethasone dipropionate 0.05% " diprolene " )

INTERVENTIONS:
Device: Ultra Violet A Device.+ Topical medical treatment — Hands of the patient are irradiated in the UVA device after soaking for 20 minutes into 10 litres of water containing psoralen "meladenine capsule".
  Arms: Phototherapy "PUVA" +traditional medical treatmentn
Device: Iontophoresis device + Topical medical treatment — Tap-water iontophoresis was given 3 times weekly for 10 min. The direct current level was slowly increased, guided by the occurrence of tingling sensations. The maximum level was 30 mA.
  Arms: Tap Water Iontophoresis + Traditional medical treatment
Drug: Topical medical treatment (Betamethasone dipropionate 0.05% " diprolene " ) — thin film of the cream is being applied to the affected areas for 2 times per day.

SUMMARY:
this study is conducted to compare the effect of phototherapy" psoralen plus UVA " bath puva to tap water iontophoresis in the treatment of atopic dermatitis in children.

DETAILED DESCRIPTION:
Sixty children were selected from the department of dermatology, Banha University Hospital. Patients were randomly assigned to (Group- A):- 20 children Patients, aged between 6-16 years old. be treated with Phototherapy, for 3 sessions per week for 8 weeks Plus the traditional medical treatment. which is the betamethasone dipropionate 0.05% " diprolene for 2 times a day for 8 weeks. (Group B): 20 children Patients, in Group-B are treated with tap water iontophoresis, for 8 weeks, 3 sessions /week: the intensity were increased according to the patient's tolerance, for 20 minutes. Plus the traditional medical treatment. (Group -C) the control group will treated by only the traditional medical treatment which is the betamethasone dipropionate 0.05% " diprolene" cream, two times a day for 8 weeks Skin thickness by ultrasonography and Patient Oriented Eczema Measure(POEM) are measured before and after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 9 to 16 years.
* Suffering from AD of dyshidrotic as well as dry types of more than 6-months duration
* Traditional types of treatment options, including oral or topical corticosteroids, proved ineffective.

Exclusion Criteria:

* Intolerance history to UV radiation.
* Skin malignancy at the area to be treated.
* Acute infection at the treated area.
* Children received radiotherapy in the area to be treated during the last 6 months.
* Children received corticosteroid therapy topically within 14 days before treatment, or systemic corticosteroids or any immunosuppressive drugs within the last 4 weeks.
* Circulatory and sensory disorders and children with diabetes mellitus.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-21 (Actual)

PRIMARY OUTCOMES:
Patient Oriented Eczema Measure" POEM" | 8 weeks of treatment
  The severity of eczema was estimated by asking young children to complete the questionnaire with the help of their parents. They were asked to leave blank any questions you feel unable to answer.

SECONDARY OUTCOMES:
Thickness of the skin " Ultrasonography" | 8 weeks of treatment
  Assessment of the skin thickness was done using the ultrasonography 7.5 MHz. The ultrasound imaging system was used to measure the thickness of the skin at the affected site

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after 6 month of publication .
Supporting Information: ICF, CSR